CLINICAL TRIAL: NCT04588506
Title: Tendon Transfer Techniques for Massive Rotator Cuff Tear Repairs: An Integrated Prospective Randomized Multicenter Trial
Brief Title: Tendon Transfer Rotator Cuff Tear
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ashfaq Hasan, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00091132
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Tears
Keywords: Massive Rotator Cuff Tears; Tendon Transfer; Rotator Cuff Tears; Tendon Transfer Techniques
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cuff tear without subscapularis tear-Lower Trapezius group (Active Comparator): Rotator cuff tears excluding the subscapularis muscle repaired using Lower Trapezius tendon
  Interventions: Procedure: Lower Trapezius Tendon Transfer Technique
- Cuff tear without subscapularis tear-Latissimus Dorsi group (Active Comparator): Rotator cuff tears excluding the subscapularis muscle repaired using Latissimus Dorsi tendon
  Interventions: Procedure: Latissimus Dorsi Tendon Transfer Technique
- Cuff tear involving subscapularis tear-Pectoralis group (Active Comparator): Rotator cuff tears involving the subscapularis muscle repaired using Pectoralis tendon
  Interventions: Procedure: Pectoralis Tendon Transfer Technique
- Cuff tear involving subscapularis tear-Latissimus Dorsi group (Active Comparator): Rotator cuff tears involving the subscapularis muscle repaired using Latissimus Dorsi tendon
  Interventions: Procedure: Latissimus Dorsi Tendon Transfer Technique

INTERVENTIONS:
Procedure: Lower Trapezius Tendon Transfer Technique — Lower Trapezius tendon used in repairing cuff tear
  Arms: Cuff tear without subscapularis tear-Lower Trapezius group
Procedure: Latissimus Dorsi Tendon Transfer Technique — Latissimus Dorsi tendon used in repairing cuff tear
  Arms: Cuff tear involving subscapularis tear-Latissimus Dorsi group; Cuff tear without subscapularis tear-Latissimus Dorsi group
Procedure: Pectoralis Tendon Transfer Technique — Pectoralis tendon used in repairing cuff tear
  Arms: Cuff tear involving subscapularis tear-Pectoralis group

SUMMARY:
This is a prospective randomized study on using muscle tendons to repair tears of the muscles on the shoulder. There are 3 muscles covering the shoulder joint- supraspinatus, infraspinatus and subscapularis. Large tears involving these muscles can be treated by using some muscle from another location of the body known as Tendon transfer techniques. These muscle tendons may be from the lower back (Latissimus Dorsi), upper pack (lower trapezius) or chest (pectoralis). There are currently no studies to show which tendon transfer technique has better outcomes.

This study comprises two trials and a total of 84 participants would be enrolled. Each trial comparing the patient reported outcomes between two tendon transfer techniques. Large tears involving the supraspinatus and infraspinatus would be repaired using either the Latissimus dorsi technique or Lower trapezius technique. 21 patients would be randomly assigned to either groups. The second trial would be comparing the Latissimus dorsi technique and pectoralis technique in large tears of the subscapularis muscle. Another 21 patients would be randomly assigned to either groups.

The investigators are studying to see if the Lower Trapezius and Pectoralis transfer techniques for muscle tear repairs would have better post-surgical outcomes compared with Latissimus Dorsi transfer technique.

For both trials, participants would be followed up for 2 years and post-surgical outcomes would be compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have massive, irreparable tear of the posterior-superior rotator cuff
* Subjects between 18 years and 65 years (≥ 18 and ≤ 65 years of age).
* Diagnosis of no to minimal glenohumeral arthritis- Hamada 1 and 2
* Subject with irreparable subscapularis tendon tear (Arms 3 and 4 ONLY)

Exclusion Criteria:

* Subjects having severe glenohumeral arthritis
* History of prior tendon transfer
* Axillary nerve injury
* Deltoid deficiency
* Subjects with pseudo paralysis
* History of post-operative deep shoulder infection
* Non-English-speaking subjects.
* Subject has any condition, that in the opinion of the investigator, would prevent them from completing this study
* Subject with irreparable subscapularis tendon tear (Arms 1 and 2 ONLY)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
12-point difference in American Shoulder and Elbow Surgeon (ASES) scores | At one year post-operative follow-up visit
  The American Shoulder and Elbow Surgeon (ASES) score is a validated and reliable outcomes measure in patients with a wide variety of shoulder disorders. The ASES questionnaire examines two domains- pain (50 points) and function (50 points)- in a self-reported questionnaire and is scored on a 100-point scale. The minimum score is zero and the maximum is 100. A higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq S Hasan, MD, Principal Investigator — U of Maryland Baltimore
Locations (1):
- U of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared